CLINICAL TRIAL: NCT07282028
Title: A Prospective, Open-label, Pivotal Study to Assess Spectacle Hearing Aid Safety and Efficacy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nuance Hearing (Industry)
Collaborators: Assuta Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 82CLD
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hearing Loss Mixed
Keywords: hearing aid; hearing disability
MeSH Terms: conditions — Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active (Experimental): Spectacle Hearing Aid
  Interventions: Device: Spectacle Hearing Aid

INTERVENTIONS:
Device: Spectacle Hearing Aid — wearing hearing aid for effectiveness assessment by hearing tests and questionnaires

SUMMARY:
Following informed consent signature and upon verification of eligibility and execution of informed consent, subjects will be assigned a study code. The study comprises two groups. Screening visit will be conducted for both groups and include hearing test battery to assess hearing aid safety and efficacy

DETAILED DESCRIPTION:
Screening Written informed consent must be obtained for each study subject prior to the commencement of the study. Upon verification of eligibility and execution of informed consent, subjects will be assigned a study code.

The study comprises two groups, stage 1 will include up to 30 participants. Stage 2 will include up to 29 participants. Stage 1 will be conducted before Stage 2, and individuals enrolled in Stage 1 will not be eligible to participate in Stage 2. The eligibility criteria for each group are outlined below.

Screening procedures include:

* ICF signature and process
* Eligibility Assessment
* Data collection: such as Age, Gender, demographic, ENT medical History
* Otoscopy performed by ENT physician
* Audiometry (Air conduction and bone conduction thresholds) might be performed as part of any other test day.
* Spectacle Hearing Aid calibration and Fitting (this activity is subjected to test with Spectacle Hearing Aid ).
* REM, aided only (optional) might be performed as part of any other test day.
* Optometrist- for glasses prescription (stage 2 only) Stage 1 :This stage involves hearing evaluation tests , which will be conducted over up to four visits, depending on participant cooperation. Each visit will be scheduled on consecutive days or up to 3 weeks apart, based on the participant's and study staff availability.

Stage 2 : After completing the screening visit, each participant will attend two additional visits. At the enrollment visit, participants will receive their Spectacle Hearing Aid along with the prescribed lenses. They will undergo training using the device and will be asked to fill out questionnaires and performed hearing tests. Additionally, the device application and Electronic Patient-Reported Outcome (ePRO) will be installed on the participants' smartphones, and a demonstration will be provided. Participants will then be required to complete the ePRO daily until the study concludes. Functional auditory test battery will be conducted. Few weeks later, participants will return to complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Perceived mild to moderate hearing loss as indicated by at least 1 positive answer to any of the signs specified by FDA: a) You have trouble hearing speech in noisy places, b) You find it hard to follow speech in groups, c) You have trouble hearing on the phone. d) Listening makes youtired, e) You need to turn up the volume on the TV or radio, and other people complain it's too loud
* Wearing corrective glasses for daily use
* Cognitive ability to understand and follow study instructions.
* The main language used in social interactions is Hebrew
* Participants must be willing to use the investigational device according to the instructions for use during the study period
* Participants must be able to use a smartphone

Exclusion Criteria:

* Hearing loss >55 dB HL
* Prior hearing aid usages for the last 12 months
* Medical history of cognitive or neurological impairment.
* Active inflammatory conditions affecting the ear
* Asymmetric or unilateral hearing loss - more than 15dB between ears in PTA4- based on screening or hearing test from the last 18 months.
* participation in stage 1 study
* Congenital ear defect or a deformed or injured ear
* In the past 6 months discharge of blood, pus or fluid
* Wax that might disturb REM test
* Sudden hearing loss in the past 6 months
* Wearer of electromagnetic medical device
* Other medical conditions/medications that would interfere with subject safety or data collection in the opinion of the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2025-07-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Spectacle Hearing Aid effectiveness | 2 weeks
  Difference in SNR-50 when performed unaided versus aided using Spectacle Hearing Aid
Spectacle Hearing Aid safety | 2 weeks
  Incidence of device or procedure related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Asssuta ramat hachayal, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
for confidentiality reasons